CLINICAL TRIAL: NCT01551927
Title: What Are the Expectations for Future Examination and Treatment in Patients Undergoing Evaluation and Treatment of Coronary Heart Disease?
Brief Title: Patients Expectations for Future Examination and Treatment
Acronym: TAPE
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: Dnr667-10; TAPE (Other: Sahlgrenska University Hospital)
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Heart Disease
Keywords: expectations
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples NtProBNP
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim: To investigate and compare women's and men's expectations before investigation and treatment of suspected coronary artery disease and to examine how these expectations are met.

Do women and men, of different ages, have the same expectations for the evaluation and treatment of stable coronary artery disease and are their expectations met in a equal degree?

Are there differences in expectations and the fulfilment of these according to age and other clinical history variables? Do the findings in the specially developed questionnaire designed to gather patients' expectations to the outcome on quality of life and degree of angina pectoris relate to their appearance in the designated forms? Is there a relationship between NTproBNP - levels, as a measure of cardiac workload, and expectations and the fulfilment of these as well as the quality of life and degree of angina pectoris?

Method: Patients will be asked to participate in the study, in the context of medical consultation before coronary angiography by a physician and / or a study nurse. This occurs during an outpatient visit at the cardiac clinic at the respective centre. Included are all patients planned for elective coronary angiography before possible revascularization during a eight month period regardless of diagnosis. Including are four hospitals in the region of Västra Götaland.

DETAILED DESCRIPTION:
Patients will be asked to participate in the study, in the context of medical consultation before coronary angiography by a physician and / or a study nurse. This occurs during an outpatient visit at the cardiac clinic at the respective centre.

Included are all patients planned for elective coronary angiography before possible revascularization during a eight month period at SKAS, NÄL, SÄS and Sahlgrenska University Hospital, this regardless of diagnosis.

Patient informed consent (attached appendix) is given to the patient before coronary angiography at the out patient visit at the cardiac clinic at the respective centre, both verbally and in writing by physician and/or nurse at the time of consultation about participation in the study. At this time the approval is signed by concerned parties. This is desired to be done only by a nurse as there is no intervention in the study. The patient has to fill out three questionnaires at two occasions (but the 10 first patients included in the reliability tests have to fill out the expectancy form a total of three times including questions about the reliability of the questionnaire). The patient also has to leave two additional blood samples.

Patients answer a questionnaire developed to measure the expectations of treatment and questionnaires measuring quality of life and presence and degree of angina pectoris, (SF-36 and SAQ Seattle Angina Questionnaire). The form of expectations is validated against the "quality of life" forms. Blood samples are taken at inclusion and again after six months and are analyzed for NTproBNP, a biochemical measure of how much strain the coronary artery disease puts on the heart muscle. We want to examine whether levels of NTproBNP before and six months after coronary angiography correlates with quality of life and expectations before the inquiry and to what extent the expectations are met. To ensure equal treatment, it is important to build a patient perspective and set offered treatment and the availability of this, in relation to the individual patient's expectations.

The following three instruments will be used to measure symptoms, functional limitation, and expectations:

* SAQ (Seattle Angina Questionnaire) is primarily formulated to measure functional status of patients with coronary artery disease. SAQ consists of 19 five-scale questions, physical limitation (nine questions), angina grade (one question), frequency of angina (two questions), satisfaction of treatment (two questions) and perception of disease (five questions), and therefore measures dimensions of physical limitations, angina degree, satisfaction of treatment and Perception of illness. The form takes about five minutes to fill in. It is not a general measurement of quality of life (7).
* SF-36 partially consists of scales measuring physical function (10 questions), role functioning-physical causes (four questions), role function-emotional reasons (three questions), social functioning (two questions) and pain (two questions), It also consists of scales for welfare, measuring mental health (five questions), vitality (four questions), general health (five questions) and change in health (one question). This instrument takes five-10 minutes to complete (8.9).
* The Expectation Form is an own developed instrument consisting of a questionnaire with 11 questions about expectations for future care and treatment, and a follow-up questionnaire six months later, to examine whether the expectations of the patient had been met. The form takes about five minutes to fill in.

The form will be evaluated and validated as follows (10):

* Reliability-test will be done by four experienced professionals, knowledgeable in the topic reviewing the questionnaire.
* The first 10 enrolled patients complete the questionnaire. This is made at an additional occasion at the time of angiography. We do a 'test re-test, with about a week apart from test to re-test. At this additional occasion patients will also answer questions about how the questionnaire was to fill in i.e. a check of the user friendliness and on how the understanding of the form was.
* Validation of the form is done with SF-36, SAQ, and NTproBNP as the criteria. All data are clinically relevant and should be recorded in the patient's medical record according to standard procedures. Case Record Form (CRF) will be coded and anonymous, and a code list will be stored at a research nurse at each, included hospital. Decoded CRF are sent to and stored at Sahlgrenska University Hospital, at the department of Cardiology. Processing and statistical data is coded and anonymous. The people managing the data are those involved in the study as well as the cardiologist research unit's coordination staff and monitoring staff.

Ethical issues must always be considered in studies where people with chronic and serious illnesses are included. Requirements for information about the study and the opportunity to connect with those responsible, respect for integrity and that none shall be harmed are fundamental ethical principles that must be followed. Anonymity and confidentiality will be guaranteed. It is also important to clarify the possibility of ending participation in the study with no consequences for further care and treatment.

Out of a privacy standpoint, there is a risk that the patient may feel exposed after filling in the questionnaire relating to life situation, personal health and the relationship with health care. We will be informing patients carefully about how we handle data and that no data may be linked to individual patients when they are compiled and presented. data is entered and managed via the Cardiology Research Unit, Sahlgrenska University Hospital. These data are available to researchers participating in the study. The lead applicant is responsible for data processing (with Statisticians) and is primarily responsible for the report.

Statistic:Data processing and statistical analysis will be done in consultation with statisticians. For about eight months, we expect, based on past experience, to be able to include 800 consecutive patients undergoing elective coronary angiography at SKAS, NÄL, SÄS and Sahlgrenska University hospital. Of these, about half is estimated to have coronary artery disease and the rest of the surveys done as part of the investigation of other cardiovascular disease as valvular disease or heart failure. The gender distribution is estimated to be about 70% men and 30% women. Dichotomous variables (baseline characteristics) are given in the frequency and compared between sexes with the chi 2 or Fisher's exact test when appropriate. Continuous variables are presented as mean values with standard deviations and compared by Student t-test. Comparisons between different age groups are made by ANOVA.

Answer from the quality of life and degree of angina pectoris instruments, converted to scores according to established schedules. Comparison of scores at baseline and six months after the angiography will be done with paired Student t-test and between groups with two-way ANOVA, or with non-parametric tests depending on the distribution of the data. The form of expectations will be analyzed to answer each question using statistics as above. The study is explorative why customary power calculation is not done. As indicated above, expected patient material will be heterogeneous with respect to clinical condition, indication for angiography, sex and age. It is therefore important to collect as many materials as possible in order to compare different groups. Based on the SF 36 it can be stated that about 50 patients in each of two groups is needed if one is to detect differences in the range of five points (total points of this instrument is often 45-50 depending on the patient group it is about) with five-point standard deviation, 0.05 and power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* <18 Years of Age.

Exclusion Criteria:

* Inability to communicate verbally or in writing.
* Unwillingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for elective coronary angiography
Sampling Method: Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grip, Prof, Principal Investigator — Sahlgrenska University Hospital Per Dubbscatan 15 41345 Göteborg Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Vastra Gotalands Regionen, Sweden

REFERENCES:
- [Background] Stables RH. Design of the 'Stent or Surgery' trial (SoS): a randomized controlled trial to compare coronary artery bypass grafting with percutaneous transluminal coronary angioplasty and primary stent implantation in patients with multi-vessel coronary artery disease. Semin Interv Cardiol. 1999 Dec;4(4):201-7. doi: 10.1006/siic.1999.0101. PMID 10738353
- [Background] Waters DD. Medical therapy versus revascularization: the atorvastatin versus revascularization treatment AVERT trial. Can J Cardiol. 2000 Jan;16 Suppl A:11A-3A. PMID 10653925
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Hambrecht R, Walther C, Mobius-Winkler S, Gielen S, Linke A, Conradi K, Erbs S, Kluge R, Kendziorra K, Sabri O, Sick P, Schuler G. Percutaneous coronary angioplasty compared with exercise training in patients with stable coronary artery disease: a randomized trial. Circulation. 2004 Mar 23;109(11):1371-8. doi: 10.1161/01.CIR.0000121360.31954.1F. Epub 2004 Mar 8. PMID 15007010
- [Background] Odell A, Grip L, Hallberg LR. Restenosis after percutaneous coronary intervention (PCI): experiences from the patients' perspective. Eur J Cardiovasc Nurs. 2006 Jun;5(2):150-7. doi: 10.1016/j.ejcnurse.2005.10.004. Epub 2005 Nov 16. PMID 16297663
- [Background] Årsrapport Swedeheart 2009 s 84 fig 76 http://www.ucr.uu.se/swedeheart/
- [Background] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Background] Sullivan M, Karlsson J. The Swedish SF-36 Health Survey III. Evaluation of criterion-based validity: results from normative population. J Clin Epidemiol. 1998 Nov;51(11):1105-13. doi: 10.1016/s0895-4356(98)00102-4. PMID 9817128
- [Background] Taft C, Karlsson J, Sullivan M. Performance of the Swedish SF-36 version 2.0. Qual Life Res. 2004 Feb;13(1):251-6. doi: 10.1023/B:QURE.0000015290.76254.a5. PMID 15058805
- [Background] Eilertsson Göran. Enkäten i praktiken. 1996,2005 www.studenlitteratur.se Studentlitteratur AB Lund 2009 sid 99-104, 151-153
- See also: Årsrapport Swedeheart 2009 s 84 fig 76 — http://www.ucr.uu.se/swedeheart/